CLINICAL TRIAL: NCT00966524
Title: Learning and Retention of Tracheal Intubation by Medical Students: Comparison of Standard Intubation Teaching Against Video-guided Intubation Teaching.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Dr François Girard, Centre Hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FG 2010-001
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Endotracheal Intubation
Keywords: Endotracheal intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video (Experimental): Teaching tracheal intubation to medical students using video-guided feedback during the procedure.
  Interventions: Procedure: Endotracheal intubation
- Standard (Active Comparator): Teaching tracheal intubation to medical students using direct visualization feedback during the procedure.
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — Pregraduates medical students will be randomized to perform endotracheal intubation with video-guided feedback (experimental arm) or endotracheal intubation using direct visualization feedback (standard technique).

SUMMARY:
Purpose: This study is designed to assess the impact of teaching tracheal intubation using video-guided feedback on the ability to perform and maintain this clinical skill by medical students.

Hypothesis: We hypothesise that, for novices, video-guided feedback provided during tracheal intubation will improve learning and retention of this clinical skill compared to standard teaching using direct visualization feedback.

DETAILED DESCRIPTION:
Introduction:

Competency in laryngoscopic tracheal intubation is a key skill to be developed during the training of medical students. Teaching this technical skill remains a challenge due to the fact that the laryngeal view is limited to one person at a time. Therefore, the feedback given during the procedure by the instructor to the student becomes limited, delayed and thus less efficient. This lack of efficiency could explain the poor success rates of tracheal intubations performed by medical students during the initial learning phase. Over the last ten years, new intubation devices incorporating optic fibers have been commercialized. These new technologies combined to video systems are now increasingly used for teaching purposes. Recent literature tends to show that this new approach could ease the learning process and increase the medical student's satisfaction towards the teaching of tracheal intubation.

Maintaining this knowledge and clinical skill can also be challenging especially for physicians who are not exposed to the intubation technique on a regular basis. Since tracheal intubation is a potentially lifesaving procedure, retention of this competency is crucial.

This study is designed to assess the impact of teaching tracheal intubation using video-guided feedback and the short and mid-term retention of the competency in a population of pregraduate medical students (clinical years 3 and 4).

Methods:

-Initial phase:

Medical students enrolled in this study will initially receive standardised training using a short video explaining the tracheal intubation technique. Then, they will be asked to intubate on mannequins for a short period of time (15 minutes).

A total of 18 medical students will be randomly assigned to the following groups:

* Group V: to perform video-guided intubations on six patients under the supervision of an anaesthesiologist.
* Group S: to perform tracheal intubation on six patients under the supervision of an anaesthesiologist using standard teaching technique (direct visualization).

Patients scheduled for elective surgery under general anaesthesia including neuromuscular blockade as part of their anaesthetic management will be considered for this study. Standard monitoring for general anaesthesia will be used. Immediately after induction of general anaesthesia, the anaesthesiologist will confirm the patient's intubation grade. Patients having an intubation grade higher than 2 on the Cormack-Lehane scale, will be excluded.

-Short-term phase (within a week from the initial phase):

Novices will be asked to perform ten tracheal intubations under the supervision of an anaesthesiologist but without any specific feedback.

-Mid-term phase (6 weeks after the initial/short-term phase):

Novices will be asked to perform ten tracheal intubations six weeks after the initial/short term phase under the supervision of an anaesthesiologist without any specific feedback. If the medical student fails to intubate the patient, the anaesthesiologist will perform the technique.

Images from all intubations will be captured on videotape for subsequent review. These images will be used to detect mucosa lacerations, oesophageal intubation, number of attempts and total time required to perform tracheal intubation.

Lastly, a questionnaire will be completed by all medical students to assess their satisfaction towards the teaching technique and their ability to perform tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Limited experience with tracheal intubation (less than 5 intubations under supervision)
* Pre-graduate medical students in their 2 clinical yea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Ease to intubate (time and number of attempts required to perform intubation) and retention of the competency (short and mid-term) | Within a week and at 6 weeks

SECONDARY OUTCOMES:
Medical students' satisfaction towards the teaching technique and their ability to perform tracheal intubation. | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: François Girard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (Hôpital Notre-Dame), Montreal, Quebec, Canada